CLINICAL TRIAL: NCT05086562
Title: Prevalence of Chronic Abdominal Pain in Migraneurs
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Principal Investigator, Magdalena S. Prüß née Volz, Principal Investigator ; PD Dr. med., Charite University, Berlin, Germany
Other Study IDs: EA1/129/21
Record Dates: First submitted 2021-09-24; First posted 2021-10-21 (Actual); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: Migraine; IBD
MeSH Terms: conditions — Migraine Disorders | interventions — Observational Studies as Topic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: observation study — observation study

SUMMARY:
To collect data on the prevalence of Chronic Abdominal Pain in Migraneurs in Germany

ELIGIBILITY:
Inclusion Criteria:

* chronic abdominal pain
* migraine

Exclusion Criteria:

* not able to sign written informed consent

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Migraneurs with Chronic Abdominal Pain
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Visual analog scale (VAS) for pain | observational, through study completion, an average of 1 year
  Number of migraneurs with chronic abdominal pain based on the VAS

CONTACTS AND LOCATIONS:
Locations (1):
- Charite University Medicine, Berlin, Germany

IPD SHARING:
Plan to Share IPD: Undecided